CLINICAL TRIAL: NCT01679860
Title: Intensive Chemo-immunotherapy as First-line Treatment in Adult Patients With Peripheral T-cell Lymphoma (PTCL)
Brief Title: Intensive Chemo-immunotherapy as First Line Treatment in Adult Patients With Peripheral T- Cell Lymphoma
Acronym: PTCL-06
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Fondazione IRCCS Istituto Nazionale dei Tumori, Milano (Other)
Responsible Party: Principal Investigator, Paolo Corradini, Director Hematology and BMT Unit, Fondazione IRCCS Istituto Nazionale dei Tumori, Milano
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PTCL-062006-004234-33
Record Dates: First submitted 2012-08-30; First posted 2012-09-06 (Estimated); Last update posted 2012-09-06 (Estimated); Status verified 2012-09

CONDITIONS: Lymphoma, T-Cell, Peripheral
MeSH Terms: conditions — Lymphoma, T-Cell, Peripheral | interventions — Alemtuzumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Clin A (Experimental): Clin A. CHOP-Campath (CHOP-C) for 2 cycles , Hyper-C-Hidam for 2 cycles and auto-SCT (stem cell transplantation) or RIC allo-SCT in advanced stage PTCL pts ≥ 18 and ≤ 60 years
  Interventions: Procedure: Clin A. CHOP-CAMPATH (Chemo-immunotherapy) + SCT
- Clin B (Experimental): Clin B: CHOP-Campath (CHOP-C) for 6 cycles . It is a combined immunochemotherapy approach in a subset of elderly pts aged > 60 ≤ 75 years
  Interventions: Drug: Clin B (CHOP- CAMPATH) Chemo-immunotherapy

INTERVENTIONS:
Procedure: Clin A. CHOP-CAMPATH (Chemo-immunotherapy) + SCT — Clin A:
  * CHOP-Campath (CHOP-C) for 2 cycles (every 21 days): Doxorubicin 50mg/m2 day +1, Vincristin 1.4mg/m2 day +1, Cyclophosphamide 750mg/m2 day +1, prednisone 100mg/m2 PO on days +1 to +5; Campath-1H (alemtuzumab) dose escalation 3-10-20mg IV days - 2, - 1, 0 (first CHOP-C) or 30mg SC day 0 (second CHOP-C). Methotrexate 12.5mg IT, Ara-C 40mg IT, Dexamethasone 4mg IT on days + 1 and 21 (first and second CHOP-C).
  * HYPER-C-HiDAM for 2 cycles: Methotrexate 1.5gr/m2 day +1; Cyclophosphamide 300mg/m2 every 12 hours days +2-3-4; ARA-C 2gr/m2 every 12 hours days +2-3-4; G-CSF 5μcg/kg/day starting from day +5 until peripheral blood stem cell harvest
  * Myeloablative regimen followed by autologous transplantation or Reduced intensity conditioning followed by allogeneic transplantation.
  Other Names: Mab - Campath (Alemtuzumab)
  Arms: Clin A
Drug: Clin B (CHOP- CAMPATH) Chemo-immunotherapy — Clin B:
  * CHOP-Campath (CHOP-C) for 6 cycles (every 21 days): Doxorubicin 50mg/m2 day +1, Vincristin 1.4mg/m2 day +1, Cyclophosphamide 750mg/m2 day +1, prednisone 100mg/m2 PO from day +1 to day +5¸ Campath-1H (alemtuzumab) 3-10mg IV on days - 1 and 0 ( first CHOP-C course) or 10mg SC on day 0 (for the following 5 C-CHOP courses). Methotrexate 12.5mg IT, Ara-C 40mg IT, Dexamethasone 4mg IT on day +1 of each CHOP-C course.
  Other Names: Mab- Campath (Alemtuzumab)
  Arms: Clin B

SUMMARY:
Peripheral T cell lymphomas (PTCL) are a rare hematologic disease. Five-year overall survival (OS) of PTCL patients (pts) ranges between 20 and 30%. Allogeneic stem cell transplantation (allo-STC) may have a curative role for these pts but its toxicity is high when myeloablative conditioning is used. Reduced intensity conditionings (RIC) can decrease transplant related toxicity and mortality. The investigators have recently proved feasibility and potential efficacy of a RIC regimen in relapsed PTCL patients.

We want to investigate whether it is possible to improve the outcome of alk negative PTCL pts, stage II-IV at diagnosis, by intensifying the therapeutic approach.

The intensification will be obtained by combining intensive chemotherapy, alemtuzumab (anti-CD52 humanised antibody) and auto- or allo-SCT in pts aged between 18 and 60 years (Clinical Study A) or adding alemtuzumab to standard chemotherapy (CHOP) in pts aged between 61 and 70 years(Clinical Study B).

DETAILED DESCRIPTION:
Inclusion criteria Clin A

* Age ≥18 < or =60 years (patients older than 60 years are excluded because of the intensive chemotherapy and transplant procedures)
* Histologically proven diagnosis of PTCL, including the following categories: PTCL-U (peripheral T-cell lymphoma, unspecified), AILD-T (angioimmunoblastic-like T-cell lymphoma), ALKneg ALCL (ALK-negative anaplastic large cell lymphoma),intestinal T - NHL
* Advanced stage disease (stage II-IV) or stage I and aaIPI score ≥ 2
* Written informed consent

Inclusion criteria Clin B

* Age >60 and ≤75 years (patients older than 75 years are excluded because of the intensive chemo-immunotherapy program)
* Histological proven diagnosis of PTCL, including the following categories: PTCL-U (peripheral T-cell lymphoma, unspecified), AILD-T (angioimmunoblastic-like T-cell lymphoma), ALKneg ALCL (ALK-negative anaplastic large cell lymphoma), intestinal T - NHL
* Advanced-stage disease (stage II-IV) or stage I and aaIPI score ≥ 2
* Informed written consent

In clinical study A (Clin A) we are planning to evaluate the efficacy and the feasibility of an intensified chemo-immunotherapy program including auto-SCT or RIC allo-SCT in advanced stage PTCL pts ≥ 18 and < or = 60 years.

In clinical study B (Clin B) we intend to verify the efficacy and the feasibility of a combined immuno-chemotherapy approach in a subset of elderly pts aged > 60 and < or = 75 years.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 <60 years (patients older than 60 years are excluded because of the intensive chemotherapy and transplant procedures)
* Histologically proven diagnosis of PTCL, including the following categories: PTCL-U (peripheral T-cell lymphoma, unspecified), AILD-T (angioimmunoblastic-like T-cell lymphoma), ALKneg ALCL (ALK-negative anaplastic large cell lymphoma),intestinal T - NHL
* Advanced stage disease (stage II-IV) or stage I and aaIPI score ≥ 2
* Written informed consent

Exclusion Criteria:

* Histological PTCL subset other than PTCL-U, AILD-T ALCL-ALKneg, intestinal T - NHL
* Central nervous system localization
* Positive serologic markers for human immunodeficiency virus (HIV), hepatitis B virus (HBV), and hepatitis C virus (HCV) infection
* Serum bilirubin levels > 2 the upper normal limit
* Clearance of creatinine < 50 ml/min
* DLCO < 50%
* Ejection fraction < 45% (or myocardial infarction in the last 12 months)
* Pregnancy or lactation
* Patient not agreeing to take adequate contraceptive measures during the study
* Psychiatric disease
* Any active, uncontrolled infection
* Type I hypersensitivity or anaphylactic reactions to proteins drugs
* Active secondary malignancy

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 92 (Actual)
Dates: Start 2006-11; Primary Completion 2011-12 (Actual); Study Completion 2012-08 (Actual)

PRIMARY OUTCOMES:
Efficacy | one year
  number of clinical responses

SECONDARY OUTCOMES:
evaluation of OS (overall survival) | 4 years
  OS time is calculated from patients enrollment to death for all causes; censored cases are pts alive at the date of last follow-up assessment.
DFS (Disease Free Survival) | 4 years
  DFS time is the interval between CR achievement and the first disease relapse or death regardless of the cause.Definition of disease response/progression will be performed according to the criteria published by Juweid et al.(J Clin Oncol. 2005; 23: 4652-61)
TRM (Treatment Related Mortality) | 4 years
  TRM will be analysed by computing the corresponding crude cumulative incidence curve, considering disease-related death as competing event.

CONTACTS AND LOCATIONS:
Overall Officials: paolo corradini, Principal Investigator — fondazione IRCCS istituto nazionale tumori Milano
Locations (17):
- Italy (17):
  - Spedali Civili di Brescia, Brescia, Brescia
  - Azienda Ospedale Vittorio Emanuele Ferrarorro S. Bambino- Università di Catania, Catania, Catania
  - Ospedale San Carlo, Potenza, Potenza
  - Azienda Ospedaliera S. Luigi, Orbassano, Torino
  - Azienda OspedalieraSan Giovanni Battista, Torino, Torino
  - Università di Torino- Azienda Ospedaliera S. Giovanni Battista, Torino, Torino
  - Policlinico Universitario Udine, Udine, Udine
  - Ospedale SS. Antonio e Biagio e Cesare Arrigo, Alessandria
  - University of Ancona - Division of Hematology, Ancona
  - Ospedale Riuniti, Bergamo - Division of Hematology, Bergamo
  - Ospedale Generale Regionale Bolzano, Bolzano
  - Ospedale S. Croce - Division of Hematology, Cuneo
  - Ospedale San Raffaele, Milano - Division of Hematology, Milan
  - Division of Hematology - Fondazione IRCCS Istituto Nazionale Tumori, Milan
  - IRCCS Ospedale Maggiore Policlinico di Milano, Milan
  - Ospedale Cervello - Bone Marrow Transplantation Unit, Palermo
  - Azienda Ospedaliera Policlinico di Verona, Verona